CLINICAL TRIAL: NCT02101281
Title: An Open-label Study Evaluating Safety and Efficacy of Recombinant Human Nerve Growth Factor (rhNGF) Eye Drops at Different Doses in Patients With Dry Eye
Brief Title: Safety and Efficacy of rhNGF Eye Drops at Different Doses in Patients With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGF0213; 2013-004271-12 (EudraCT Number)
Record Dates: First submitted 2014-03-20; First posted 2014-04-02 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — cenegermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - rhNGF 20 μg/mL (Experimental): (first planned dose): drop (35 μL) corresponding to 0.70 μg of rhNGF (recombinant human Nerve Growth Factor) was instilled into each eye twice a day (b.i.d.) every 12±2 h for a total daily dose of 2.8 μg (both eyes), for 28 consecutive days. The total dose was 78.4 μg/28 days.
  Interventions: Drug: rhNGF 20 µg/mL
- Group 2 - rhNGF 4 μg/mL (Experimental): after completion of Group 1 treatment, one drop (35 μL) corresponding to 0.14 μg of rhNGF (recombinant human Nerve Growth Factor) instilled into each eye b.i.d. every 12±2 h for a total daily dose of 0.56 μg, for 28 consecutive days. Total dose was 15.68 μg/28 days.
  Interventions: Drug: rhNGF 4 µg/mL

INTERVENTIONS:
Drug: rhNGF 20 µg/mL — 1 drop for each eye, twice daily for 28 day
  Other Names: cenegermin, recombinant human Nerve Growth Factor
  Arms: Group 1 - rhNGF 20 μg/mL
Drug: rhNGF 4 µg/mL — 1 drop each eye, twice daily for 28 day
  Other Names: cenegermin, recombinant human Nerve Growth Factor
  Arms: Group 2 - rhNGF 4 μg/mL

SUMMARY:
The primary objective of this study was to assess the efficacy and safety of different doses of rhNGF when administered as eye drops to patients with dry eye.

DETAILED DESCRIPTION:
This is an open-label study evaluating safety and efficacy of recombinant human nerve growth factor (rhNGF) eye drops at different doses in patients with Dry Eye

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 18 years old;
2. Required use of artificial tears for the treatment of Dry Eye within the 3 months prior to study enrolment;
3. Current use or recommended use of artificial tears for the treatment of Dry Eye;
4. Average VAS score for typical symptoms of Dry Eye (foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia) ≥ 25 mm;
5. Corneal staining score with lissamine green > 3 using the NEI corneal grading system in the worse eye (study eye);
6. Conjunctival staining score > 3 using the NEI conjunctival grading system in the worse eye (study eye);
7. Schirmer test without anaesthesia ≤ 10 mm/5 minutes in the worse eye (study eye);
8. Tear film break-up time (TBUT) ≤ 10 seconds in the worse eye (study eye);
9. A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period

Exclusion Criteria:

1. Patient not suitable to participate in the study in the opinion of the investigator;
2. Patient with a mild or moderate Dry Eye condition (severity level less than 3 according to the Report of the International Dry Eye Workshop -DEWS, 2007) if fourteen (14) patients with mild or moderate dry eye condition have been already enrolled in the current treatment group (Group 1 and Group 2 separately);
3. Patient has had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or has a clinically significant allergy to drugs, foods, amide local anaesthetics or other materials including commercial artificial tears containing Hypromellose (in the opinion of the investigator);
4. Use of topical cyclosporine, topical corticosteroids or any other topical medication for the treatment of dry eye in either eye within 30 days of study enrolment. Use of own artificial tears is allowed until Visit 2;
5. Any ocular disease other than Dry Eye requiring treatment with topical medications in either eye within 30 days of study enrolment;
6. Any active ocular infection or active inflammation in either eye unrelated to Dry Eye;
7. Presence or history of any systemic or ocular disorder, condition or disease that could possibly interfere with the conduct of the required study procedures or the interpretation of the study results;
8. Use of therapeutic or Refractive Contact lenses in either eye within 30 days of study enrolment;
9. History of ocular surgery in the study eye, including corneal refractive procedures, within 90 days of study enrolment;
10. Participation in another clinical study at the same time as the present and within 30 days of study enrolment;
11. History of drug, medication or alcohol abuse or addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Medical University of Vienna, Vienna General Hospital, AKH
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Sacchetti M, Lambiase A, Schmidl D, Schmetterer L, Ferrari M, Mantelli F, Allegretti M, Garhoefer G. Effect of recombinant human nerve growth factor eye drops in patients with dry eye: a phase IIa, open label, multiple-dose study. Br J Ophthalmol. 2020 Jan;104(1):127-135. doi: 10.1136/bjophthalmol-2018-312470. Epub 2019 Apr 3. PMID 30944103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The investigator included in the study 40 subjects. After inclusion, all the 40 subjects took the study treatment. In detail, the first 20 enrolled subjects received rhNGF 20 μg/mL eye drops (Group 1) and the last 20 enrolled subjects received rhNGF 4 μg/mL eye drops (Group 2).
Groups:
- Group 1 - rhNGF 20 μg/mL: (first planned dose): one drop (35 μL) corresponding to 0.70 μg of rhNGF was instilled into each eye twice a day (b.i.d.) every 12±2 h for a total daily dose of 2.8 μg (both eyes), for 28 consecutive days. Total dose was 78.4 μg/28 days.
  rhNGF 20 µg/mL: 1 drop for each eye, twice daily for 28 day
- Group 2 - rhNGF 4 μg/mL: after completion of Group 1 treatment, one drop (35 μL) corresponding to 0.14 μg of rhNGF was instilled into each eye b.i.d. every 12±2 h for a total daily dose of 0.56 μg, for 28 consecutive days. Total dose was 15.68 μg/28 days.
  rhNGF 4 µg/mL: 1 drop each eye, twice daily for 28 day
Period: Overall Study
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set: all enrolled patients, who received at least one dose of the IMP.
  This analysis set was used for the efficacy analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (12.0) | 55.9 (14.8) | 52.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Austria | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Frequency of Dry Eye Symptoms (SANDE)
Description: The SANDE is a short questionnaire to evaluate the frequency of ocular dryness and/or irritation symptoms. For the assessment, the patients mark on a 100 mm Visual Analogue Scale (VAS) line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks. The SANDE scores (0-100) will be then evaluated for frequency per day.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: FAS subjects: all enrolled patients, who received at least one dose of the IMP. This analysis set was used for the efficacy analysis
Measure: Mean (Standard Deviation); unit: Frequency of symptoms per day
Groups:
- SANDE Changes From Baseline With rhNGF 20 μg/mL: Mean (±SD) changes from baseline and the outcome of their comparison with baseline after treatment with rhNGF 20 μg/mL - Day 1, 8, 29, 56
- SANDE Changes From Baseline With rhNGF 4 μg/mL: Mean (±SD) changes from baseline and the outcome of their comparison with baseline after treatment with rhNGF 4 μg/mL - Day 1, 8, 29, 56
Arm/Group | SANDE Changes From Baseline With rhNGF 20 μg/mL | SANDE Changes From Baseline With rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
Frequency of symptoms per day
  Day 1 | -8.0 (15.9) | -10.0 (24.8)
  Day 8 | -15.0 (20.1) | -23.4 (26.0)
  Day 29 | -26.9 (24.5) | -24.5 (22.2)
  Day 56 | -30.1 (18.3) | -28.0 (23.6)

2. Primary Outcome: Change From Baseline in Severity of Dry Eye Symptoms (SANDE)
Description: The SANDE is a short questionnaire to evaluate the severity of ocular dryness and/or irritation symptoms. For the assessment, the patients mark on the 100 mm VAS line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left-hand end of the line to the point that the patient marks. The SANDE scores (0-100) will be then evaluated for severity. The higher the score, the worse the outcome.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SANDE Changes From Baseline With rhNGF 20 μg/mL | SANDE Changes From Baseline With rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
units on a scale
  Day 1 | -7.6 (20.1) | -9.9 (21.9)
  Day 8 | -11.7 (19.9) | -21.1 (29.6)
  Day 29 | -27.0 (28.4) | -28.9 (28.4)
  Day 56 | -29.0 (23.9) | -28.2 (26.9)

3. Primary Outcome: Change From Baseline in Ocular Surface Vital Staining (National Eye Institute [NEI] Scale)
Description: The cornea is divided into five sectors (central, superior, inferior, nasal and temporal), each of which is scored on a scale of 0-3, with a maximal score of 15. Both nasally and temporally, the conjunctiva is divided into a superior paralimbal area, an inferior paralimbal area and a peripheral area with a grading scale of 0-3 and with a maximal score of 9 for the nasal and temporal conjunctiva.
  Staining was derived as the sum of scores in the various sectors. The higher the total score the more compromised is the ocular surface.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ocular Surface Staining With LG With rhNGF 20 μg/mL; Ocular Surface Staining With LG With rhNGF 4 μg/mL: Mean (±SD) changes from baseline and the outcome of their comparison with baseline after treatment with rhNGF 20 μg/mL - Day 1, 8, 29, 56
Arm/Group | Ocular Surface Staining With LG With rhNGF 20 μg/mL | Ocular Surface Staining With LG With rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
units on a scale
  Central cornea, Day 1 vs Day -15 | -0.1 (0.8) | 0.0 (0.0)
  Central cornea, Day 8 vs Day -15 | -0.4 (0.9) | -0.2 (0.5)
  Central cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Central cornea, Day 29 vs Day -15 | -0.7 (0.9) | -0.3 (0.7)
  Central cornea, Day 56 vs Day -15 | -0.8 (0.9) | -0.4 (0.9)
  Superior cornea, Day 1 vs Day -15 | 0.2 (0.4) | -0.1 (0.2)
  Superior cornea, Day 8 vs Day -15 | -0.2 (0.7) | -0.1 (0.7)
  Superior cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Superior cornea, Day 29 vs Day -15 | -0.4 (0.5) | -0.3 (1.1)
  Superior cornea, Day 56 vs Day -15 | -0.3 (0.6) | -0.5 (0.8)
  Inferior cornea, Day 1 vs Day -15 | -0.2 (0.7) | -0.2 (0.5)
  Inferior cornea, Day 8 vs Day -15 | -0.6 (0.7) | -0.5 (0.5)
  Inferior cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Inferior cornea, Day 29 vs Day -15 | -1.2 (0.5) | -0.9 (0.8)
  Inferior cornea, Day 56 vs Day -15 | -1.1 (0.5) | -0.9 (0.9)
  Nasal cornea, Day 1 vs Day -15 | -0.1 (0.6) | 0.0 (0.3)
  Nasal cornea, Day 8 vs Day -15 | -0.7 (0.5) | -0.2 (0.5)
  Nasal cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Nasal cornea, Day 29 vs Day -15 | -1.0 (0.5) | -0.7 (0.6)
  Nasal cornea, Day 56 vs Day -15 | -1.0 (0.7) | -0.5 (0.7)
  Temporal cornea, Day 1 vs Day -15 | -0.3 (1) | 0.0 (0.3)
  Temporal cornea, Day 8 vs Day -15 | -0.9 (0.7) | -0.3 (0.6)
  Temporal cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Temporal cornea, Day 29 vs Day -15 | -0.8 (0.6) | -0.6 (0.6)
  Temporal cornea, Day 56 vs Day -15 | -1.0 (0.6) | -0.6 (0.8)
  Total score cornea, Day 1 vs Day -15 | -0.4 (2.4) | -0.2 (0.8)
  Total score cornea, Day 8 vs Day -15 | -2.7 (1.7) | -1.2 (1.4)
  Total score cornea, Day 29 vs Day -15 | -4.0 (1.5) | -2.9 (1.7)
  Total score cornea, Day 56 vs Day -15: number analyzed (Participants) | 20 | 19
  Total score cornea, Day 56 vs Day -15 | -4.0 (1.7) | -0.9 (2.5)
  Day 1 - Superior Paralimbal Nasal Conjunctiva | -0.3 (0.4) | 0.0 (0.5)
  Day 8 - Superior Paralimbal Nasal Conjunctiva | -0.4 (0.9) | -0.3 (0.6)
  Day 29 - Superior Paralimbal Nasal Conjunctiva: number analyzed (Participants) | 20 | 19
  Day 29 - Superior Paralimbal Nasal Conjunctiva | -0.9 (1.1) | -0.4 (0.6)
  Day 56 - Superior Paralimbal Nasal Conjunctiva | -0.6 (0.9) | -0.5 (0.6)
  Day 1 - Inferior Paralimbal Nasal Conjunctiva | -0.2 (0.7) | 0.1 (0.4)
  Day 8 - Inferior Paralimbal Nasal Conjunctiva | -0.5 (0.8) | -0.4 (0.6)
  Day 29 - Inferior Paralimbal Nasal Conjunctiva: number analyzed (Participants) | 20 | 19
  Day 29 - Inferior Paralimbal Nasal Conjunctiva | -0.9 (0.7) | -0.4 (0.5)
  Day 56 - Inferior Paralimbal Nasal Conjunctiva | -0.5 (0.7) | -0.3 (0.6)
  Peripheral Nasal Conjunctiva, Day 1 vs Day -15 | 0.0 (0.9) | 0.2 (0.6)
  Peripheral Nasal Conjunctiva, Day 8 vs Day -15 | -0.5 (1.1) | -0.4 (0.7)
  Peripheral Nasal Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Peripheral Nasal Conjunctiva, Day 29 vs Day -15 | -1.0 (0.8) | -0.5 (0.8)
  Peripheral Nasal Conjunctiva, Day 56 vs Day -15 | -0.7 (1.0) | -0.7 (0.8)
  Day 1 - Superior Paralimbal Temporal Conjunctiva | -0.2 (0.7) | 0.1 (0.3)
  Day 8 - Superior Paralimbal Temporal Conjunctiva | -0.5 (0.8) | -0.1 (0.7)
  Day 29 - Superior Paralimbal Temporal Conjunctiva: number analyzed (Participants) | 20 | 19
  Day 29 - Superior Paralimbal Temporal Conjunctiva | -0.9 (0.8) | -0.4 (0.8)
  Day 56 - Superior Paralimbal Temporal Conjunctiva | -0.6 (0.9) | -0.5 (0.7)
  Day 1 - Inferior Paralimbal Temporal Conjunctiva | -0.3 (0.6) | 0.2 (0.5)
  Day 8 - Inferior Paralimbal Temporal Conjunctiva | -0.6 (0.9) | 0.0 (0.5)
  Day 29 - Inferior Paralimbal Temporal Conjunctiva: number analyzed (Participants) | 20 | 19
  Day 29 - Inferior Paralimbal Temporal Conjunctiva | -1.0 (0.8) | -0.2 (0.7)
  Day 56 - Inferior Paralimbal Temporal Conjunctiva | -0.8 (1.0) | -0.1 (0.8)
  Peripheral Temporal Conjunctiva, Day 1 vs Day -15 | -0.4 (0.7) | 0.0 (0.6)
  Peripheral Temporal Conjunctiva, Day 8 vs Day -15 | -0.9 (0.6) | 0.0 (0.8)
  Peripheral Temporal Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Peripheral Temporal Conjunctiva, Day 29 vs Day -15 | -1.1 (0.9) | -0.2 (0.8)
  Peripheral Temporal Conjunctiva, Day 56 vs Day -15 | -0.7 (1.0) | -0.2 (0.8)
  Total Score Conjunctiva, Day 1 vs Day -15 | -1.2 (2.5) | 0.5 (1.4)
  Total Score Conjunctiva, Day 8 vs Day -15 | -3.3 (2.9) | -1.1 (1.8)
  Total Score Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Total Score Conjunctiva, Day 29 vs Day -15 | -5.6 (3.2) | -2.2 (1.8)
  Total Score Conjunctiva, Day 56 vs Day -15 | -3.9 (3.3) | -2.2 (2.0)

4. Primary Outcome: Change From Baseline in Tear Wetting Distance as Determined by Schirmer Tear Test I - Study Eye
Description: The Schirmer test type I (without anaesthesia) was performed to measure aqueous tear secretion prior to the instillation of any dilating or anaesthetic eye drops. The rounded tip of a standardized paper strip is inserted into the lower fornix of the eye, and the wetted length extending out from the lower lid is recorded after 5 min of eye closure. Both eyes could be tested at the same time. Changes from baseline in values of Schirmer's test type I are summarised by eye and evaluation visit, and stratified by severity level. The longer the wetted length the healthier the status of the eye. Only study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: FAS subjects:
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Schirmer's Test Type I Changes From Baseline - rhNGF 20 μg/mL: Mean (±SD) changes from baseline and the outcome of their comparison with baseline after treatment with rhNGF 20 μg/mL - Day 1, 8, 29, 56
- Schirmer's Test Type I Changes From Baseline - rhNGF 4 μg/mL: Mean (±SD) changes from baseline and the outcome of their comparison with baseline after treatment with rhNGF 4 μg/mL - Day 1, 8, 29, 56
Arm/Group | Schirmer's Test Type I Changes From Baseline - rhNGF 20 μg/mL | Schirmer's Test Type I Changes From Baseline - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
millimeters
  Day 1 vs Day -15: number analyzed (Participants) | 20 | 13
  Day 1 vs Day -15 | 1.3 (4.9) | 1.4 (5.2)
  Day 8 vs Day -15: number analyzed (Participants) | 20 | 13
  Day 8 vs Day -15 | 4.5 (7.2) | 0.8 (5.6)
  Day 29 vs Day -15: number analyzed (Participants) | 20 | 12
  Day 29 vs Day -15 | 5.3 (6.5) | 3.2 (6.0)
  Day 56 vs Day -15: number analyzed (Participants) | 20 | 13
  Day 56 vs Day -15 | 4.6 (8.3) | 4.6 (6.7)

5. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs),
Description: The treatment-emergent adverse events were recorded throughout the whole study.
Time Frame: Throughout the study up to day 56
Population: Safety set: all patients who received at least one dose of the IMP. This analysis set was used for the safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
Participants | 14 | 15

6. Secondary Outcome: Change From Baseline in Ocular Tolerability (Visual Analogue Scale, VAS)
Description: A ocular tolerability score was determined using a 100 mm VAS on which 0 meant No symptoms and 100 meant the Worst possible discomfort. The patients subjectively evaluated their ocular symptoms (foreign body sensation, burning or stinging, itching, pain, sticky feeling, blurred vision and photophobia) using the VAS giving the value they were feeling from none to an extreme value.
  The ocular symptoms were evaluated by the patients through the scale. Only the study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: FAS: all enrolled patients, who received at least one dose of the IMP. This analysis set was used for the efficacy analysis
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
Units on a scale
  Foreign Body Sensation, Day 1 vs Day -15 | -18.4 (18.6) | -1.2 (22.8)
  Foreign Body Sensation, Day 8 vs Day -15 | -25.2 (19.4) | -19.9 (24.0)
  Foreign Body Sensation, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Foreign Body Sensation, Day 29 vs Day -15 | -31.4 (24.3) | -30.4 (33.5)
  Foreign Body Sensation, Day 56 vs Day -15 | -30.7 (20.5) | -29.9 (28.2)
  Burning/Stinging, Day 1vs Day -15 | -21.3 (21.1) | -7.4 (17.3)
  Burning/Stinging, Day 8 vs Day -15 | -25.9 (21.1) | -13.7 (30.9)
  Burning/Stinging, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Burning/Stinging, Day 29 vs Day -15 | -32.7 (21.8) | -24.1 (30.9)
  Burning/Stinging, Day 56 vs Day -15 | -30.2 (19.6) | -29.9 (28.1)
  Itching, Day 1 vs Day -15 | -14.6 (20.4) | -14.0 (22.3)
  Itching, Day 8 vs Day -15 | -23.8 (18.2) | -24.1 (29.6)
  Itching, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Itching, Day 29 vs Day -15 | -30.7 (20.3) | -33.9 (32.8)
  Itching, Day 56 vs Day -15 | -26.0 (25.8) | -35.2 (33.0)
  Pain - Day 1 vs Day -15 | -19.2 (21.6) | -2.5 (14.9)
  Pain, Day 8 vs Day -15 | -15.4 (30.0) | -4.1 (29.8)
  Pain, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Pain, Day 29 vs Day -15 | -24.4 (21.7) | -14.9 (28.9)
  Pain, Day 56 vs Day -15 | -24.9 (20.1) | -16.9 (22.6)
  Sticky feeling, Day 1 vs Day -15 | -9.2 (15.1) | -1.4 (26.0)
  Sticky feeling, Day 8 vs Day -15 | -11.7 (20.0) | -16.9 (27.1)
  Sticky feeling, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Sticky feeling, Day 29 vs Day -15 | -12.7 (22.1) | -22.7 (23.8)
  Sticky feeling, Day 56 vs Day -15 | -13.2 (22.0) | -22.6 (22.5)
  Blurred vision, Day 1 vs Day -15 | -24.0 (21.1) | -7.0 (17.6)
  Blurred vision, Day 8 vs Day -15 | -29.9 (30.7) | -17.2 (25.9)
  Blurred vision, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Blurred vision, Day 29 vs Day -15 | -41.0 (28.4) | -31.6 (28.3)
  Blurred vision, Day 56 vs Day -15 | -39.4 (27.4) | -28.4 (27.2)
  Photophobia, Day 1 vs Day -15 | -21.0 (23.1) | 5.0 (23.9)
  Photophobia, Day 8 vs Day -15 | -27.1 (22.8) | -10.8 (35.9)
  Photophobia, Day 29 vs Day -15 | -31.5 (22.6) | -20.8 (42.8)
  Photophobia, Day 56 vs Day -15 | -32.3 (21.9) | -23.1 (29.8)

7. Secondary Outcome: Change From Baseline in Slit Lamp Examination
Description: SLE grading of the eyelids, lashes, conjunctiva, cornea, lens, iris and anterior chamber was done according to the following scales:
  Eyelid - Meibomian glands (evaluation of the central ten Meibomian gland openings in the mid-portion of the upper eyelid):
  0, 1, 2, 3 = None, Mild, Moderate, Severe gland plugging Eyelid - Erythema 0, 1, 2, 3,4 = None, Mild, Moderate, Severe, Very severe redness of lid margin and/or skin Eyelid - Oedema 0, 1, 2, 3,4 = None, Mild, Moderate, Severe, Very severe oedema Lashes 0 = Normal
  1 = Abnormal Conjunctiva - Erythema 0, 1, 2, 3, 4 = None, Mild, Moderate, Severe erythema Conjunctiva - Oedema 0, 1, 2, 3, 4 = None, Mild, Moderate, Severe, Very severe swelling Lens 0, 1, 2, 3 = No, Mild, Moderate, Severe opacification N/A = Patient with artificial lens Iris 0 = Normal
  1 = Abnormal. Anterior Chamber Inflammation 0, 1, 2, 3, = No, Mild, Moderate, Severe, Very severe Tyndall effect
  Only the study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Da 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
units on a scale
  Eyelid - Meibomian glands, Day 1 vs Day -15 | 0.1 (0.6) | -0.2 (0.4)
  Eyelid - Meibomian glands, Day 8 vs Day -15 | -0.1 (0.6) | -0.3 (0.6)
  Eyelid - Meibomian glands, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Eyelid - Meibomian glands, Day 29 vs Day -15 | -0.6 (0.8) | -0.3 (0.7)
  Eyelid - Meibomian glands, Day 56 vs Day -15 | -0.4 (0.9) | -0.3 (0.7)
  Eyelid - erythema, Day 1 vs Day -15 | -0.1 (0.6) | -0.1 (0.2)
  Eyelid - erythema, Day 8 vs Day -15 | -0.3 (0.7) | 0.0 (0.6)
  Eyelid - erythema, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Eyelid - erythema, Day 29 vs Day -15 | -0.8 (0.6) | 0.1 (0.7)
  Eyelid - erythema, Day 56 vs Day -15 | -0.8 (0.7) | -0.1 (0.6)
  Eyelid - Oedema, Day 1 vs Day -15 | 0.2 (0.5) | 0.0 (0.3)
  Eyelid - Oedema, Day 8 vs Day -15 | -0.2 (0.5) | 0.2 (0.5)
  Eyelid - Oedema, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Eyelid - Oedema, Day 29 vs Day -15 | -0.4 (0.5) | 0.2 (0.6)
  Eyelid - Oedema, Day 56 vs Day -15 | -0.4 (0.5) | 0.0 (0.6)
  Lashes, Day 1 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Lashes, Day 8 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Lashes, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Lashes, Day 29 vs Day -15 | 0.0 (0.0) | -0.3 (0.7)
  Lashes, Day 56 vs Day -15 | 0.0 (0.0) | -0.3 (0.8)
  Conjunctiva - Erythema, Day 1 vs Day -15 | -0.2 (0.5) | -0.3 (0.6)
  Conjunctiva - Erythema, Day 8 vs Day -15 | -0.4 (0.7) | -0.4 (0.7)
  Conjunctiva - Erythema, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Conjunctiva - Erythema, Day 29 vs Day -15 | -0.5 (0.7) | -0.4 (0.9)
  Conjunctiva - Erythema, Day 56 vs Day -15 | -0.5 (0.9) | -0.6 (1.0)
  Conjunctiva - Oedema, Day 1 vs Day -15: number analyzed (Participants) | 20 | 19
  Conjunctiva - Oedema, Day 1 vs Day -15 | 0.0 (0.6) | -0.3 (0.6)
  Conjunctiva - Oedema, Day 8 vs Day -15 | -0.4 (0.8) | -0.4 (0.7)
  Conjunctiva - Oedema, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Conjunctiva - Oedema, Day 29 vs Day -15 | -0.7 (0.9) | -0.4 (0.9)
  Conjunctiva - Oedema, Day 56 vs Day -15 | -0.3 (1.0) | -0.6 (1.0)
  Lens, Day 1 vs Day -15: number analyzed (Participants) | 19 | 16
  Lens, Day 1 vs Day -15 | 0.1 (0.2) | 0.0 (0.0)
  Lens, Day 8 vs Day -15: number analyzed (Participants) | 19 | 16
  Lens, Day 8 vs Day -15 | 0.0 (0.3) | 0.0 (0.0)
  Lens, Day 29 vs Day -15: number analyzed (Participants) | 19 | 15
  Lens, Day 29 vs Day -15 | -0.1 (0.5) | -0.1 (0.3)
  Lens, Day 56 vs Day -15: number analyzed (Participants) | 19 | 16
  Lens, Day 56 vs Day -15 | -0.1 (0.5) | -0.1 (0.3)
  Iris, Day 1 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Iris, Day 8 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Iris, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Iris, Day 29 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Iris, Day 56 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Anterior Chamber Inflammation, Day 1 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Anterior Chamber Inflammation, Day 8 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Anterior Chamber Inflammation, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Anterior Chamber Inflammation, Day 29 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)
  Anterior Chamber Inflammation, Day 56 vs Day -15 | 0.0 (0.0) | 0.0 (0.0)

8. Secondary Outcome: Change From Baseline in Tear Wetting Distance as Determined by Schirmer Tear Test II - Study Eye
Description: The Schirmer test type II (with anaesthesia) was performed to measure aqueous tear secretion following the instillation of a preservative-free anaesthetic eye drop (Oxybuprocaine Chlorhydrate 0.4%). The rounded tip of a standardized paper strip is inserted into the lower fornix of the eye, and the wetted length extending out from the lower lid is recorded after 5 min of eye closure. Both eyes could be tested at the same time. Changes from baseline in values of Schirmer's test type I are summarised by eye and evaluation visit and stratified by severity level. The longer the wetted length the healthier the status of the eye. Only study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
millimeters
  Day 1 vs Day -15 | -2.0 (9.5) | 2.5 (5.7)
  Day 8 vs Day -15 | 1.6 (13.3) | 2.1 (5.9)
  Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Day 29 vs Day -15 | 3.8 (8.7) | 6.5 (8.9)
  Day 56 vs Day -15 | 2.2 (11.4) | 6.9 (5.7)

9. Secondary Outcome: Change From Baseline in Tear Film Break-Up Time (TFBUT)
Description: TFBUT was measured by determining the time to tear break-up. The TFBUT was performed after instillation of 5 μl of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. With the aid of a slit lamp at 10X magnification using cobalt blue illumination, the examiner will monitor the integrity of the tear film, noting the time it takes to form lacunae (clear spaces in the tear film) from the time that the eye is opened after the last blink. The longer the time the better the integrity of the tear film.
  Only Study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
seconds
  Average Tear Film Break-Up Time, Day 1 vs Day -15 | 0.6 (2.1) | -0.7 (1.7)
  Average Tear Film Break-Up Time, Day 8 vs Day -15 | 1.5 (2.6) | -0.3 (2.1)
  Average Tear Film Break-Up Time, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Average Tear Film Break-Up Time, Day 29 vs Day -15 | 2.6 (2.9) | -0.6 (2.2)
  Average Tear Film Break-Up Time, Day 56 vs Day -15 | 2.2 (2.8) | -0.3 (2.8)

10. Secondary Outcome: Change From Baseline in Corneal Fluorescein Staining
Description: Fluorescein staining of the cornea is a methodology to visualize corneal epithelial defects under slit lamp microscopy in patients with suspicious or known Dry Eye Disease (DED). Fluorescein dyed - impregnated paper strips were used. Before placing the strip in the lower fornix of the eye, a drop of sterile saline was added to the strip.
  The cornea was divided into five sectors (central, superior, inferior, nasal and temporal), each of which was scored on a scale of 0-3, with a maximal global score of 15.
  For a better reading under the slit lamp, no intense illumination beam was used, since it could reduce the contrast and lead to an underestimation of grading.
  The lower the score the lower the corneal damage.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
units on a scale
  Central cornea, Day 1 vs Day -15 | -0.1 (0.5) | 0.1 (0.3)
  Central cornea, Day 8 vs Day -15 | -0.3 (0.9) | -0.2 (0.5)
  Central cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Central cornea, Day 29 vs Day -15 | -0.5 (0.8) | -0.2 (0.7)
  Central cornea, Day 56 vs Day -15 | -0.5 (0.7) | -0.1 (0.9)
  Superior cornea, Day 1 vs Day -15 | 0.1 (0.9) | 0.1 (0.5)
  Superior cornea, Day 8 vs Day -15 | -0.4 (0.8) | -0.1 (0.7)
  Superior cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Superior cornea, Day 29 vs Day -15 | -0.4 (0.8) | -0.1 (0.9)
  Superior cornea, Day 56 vs Day -15 | -0.1 (0.8) | -0.4 (0.8)
  Inferior cornea, Day 1 vs Day -15 | -0.1 (0.6) | 0.1 (0.4)
  Inferior cornea, Day 8 vs Day -15 | -0.4 (0.8) | -0.1 (0.6)
  Inferior cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Inferior cornea, Day 29 vs Day -15 | -0.8 (0.9) | -0.3 (1.0)
  Inferior cornea, Day 56 vs Day -15n | -0.8 (1.0) | -0.3 (0.9)
  Nasal cornea, Day 1 vs Day -15 | -0.2 (0.6) | 0.1 (0.7)
  Nasal cornea, Day 8 vs Day -15 | -0.5 (0.8) | 0.0 (0.8)
  Nasal cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Nasal cornea, Day 29 vs Day -15 | -0.9 (0.9) | -0.3 (0.9)
  Nasal cornea, Day 56 vs Day -15 | -0.8 (0.8) | -0.2 (0.5)
  Temporal cornea, Day 1 vs Day -15 | 0.0 (0.6) | 0.1 (0.6)
  Temporal cornea, Day 8 vs Day -15 | -0.4 (0.8) | -0.1 (0.8)
  temporal cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  temporal cornea, Day 29 vs Day -15 | -0.6 (0.7) | -0.4 (0.8)
  Temporal cornea, Day 56 vs Day -15 | -0.8 (0.7) | -0.3 (0.8)
  Total score cornea, Day 1 vs Day -15 | -0.3 (2.6) | 0.4 (1.4)
  Total score cornea, Day 8 vs Day -15 | -1.9 (3.0) | -0.4 (2.2)
  Total score cornea, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Total score cornea, Day 29 vs Day -15 | -3.1 (2.7) | -1.2 (2.9)
  Total score cornea, Day 56 vs Day -15 | -2.9 (2.7) | -1.2 (2.8)

11. Secondary Outcome: Change From Baseline in Corneal Sensitivity to Contact (Cochet-Bonnet Aesthesiometry)
Description: Corneal sensitivity was measured in cm through the Luneau-Cochet-Bonnet aesthesiometer. This contains a thin, retractable, nylon monofilament that extends up to 6 cm in length. Variable pressure can be applied to the cornea by adjusting the monofilament length. The monofilament length ranges from 6 to 0.5 cm. As the monofilament length is decreased the pressure increases from 11 mm/g to 200 mm/g. The filament is retracted incrementally in 0.5 cm until the patient gives a positive reaction indicating that the contact of the monofilament on the cornea has been sensed. The shorter filament lengths indicate decreased corneal sensation. The length of the filament (in cm) at which the patient sensed the contact with the cornea is recorded.
  Only study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
cm
  Filament Length of Contact Sensation,Day1vsDay-15 | 0.05 (0.58) | 0.20 (0.41)
  Filament Length of Contact Sensation,Day8vsDay-15 | 0.03 (0.41) | 0.38 (0.94)
  Filament Length of Contact Sensation,Day29vsDay-15: number analyzed (Participants) | 20 | 19
  Filament Length of Contact Sensation,Day29vsDay-15 | 0.33 (0.82) | 0.39 (1.25)
  Filament Length of Contact Sensation,Day56vsDay-15 | 0.28 (0.60) | 0.50 (1.19)

12. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: IOP was performed using either Goldmann applanation tonometry or a handheld applanation tonometer (e.g. Tonopen) after the instillation of a topical anaesthetic. IOP was measured in both eyes after completion of all other slit lamp examinations to avoid potential interference with the other evaluations. Only study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
mmHg
  Day 1 vs Day -15 | -0.9 (1.6) | 0.2 (2.3)
  Day 8 vs Day -15 | -1.9 (2.2) | 0.5 (3.2)
  Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Day 29 vs Day -15 | -1.6 (2.6) | 1.3 (3.1)
  Day 56 vs Day -15 | -1.7 (3.0) | 0.9 (2.9)

13. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI)
Description: The OSDI is based on a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning. The 12 items of the OSDI questionnaire are graded on a 0-4 scale as follows:
  Grade 0 = none Grade 1 = some Grade 2 = half Grade 3 = most Grade 4 = all
  The total OSDI score was then calculated on the basis of the following formula:
  OSDI=[(sum of scores for all questions answered) × 100]/[(total number of questions answered) × 4].
  Thus, the OSDI total score scales from 0 to 100, with higher scores representing greater disability.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
score on a scale
  Day 1 vs Day -15 | -5.37 (9.38) | -0.22 (12.90)
  Day 8 vs Day -15 | -14.33 (13.03) | -10.39 (16.88)
  Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Day 29 vs Day -15 | -22.92 (18.73) | -18.75 (24.78)
  Day 56 vs Day -15 | -23.47 (22.72) | -14.76 (17.91)

14. Secondary Outcome: Change From Baseline in Visual Acuity (BCDVA)
Description: Values of Best-Corrected Distance Visual Acuity (BCDVA) scores were measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) score. The ETDRS charts use letters, or a geometric progression in letter size from line to line, under standardized lighting conditions. The patient starts at the top of the chart, or on the last row where he or she can read all of the letters, and reads down the chart until he or she reaches a row where a minimum of three letters on a line cannot be read. The patient is scored by how many letters could be correctly identified. Therefore, the higher the number of letters the higher the visual acuity.
  Changes in the ETDRS score from baseline (screening visit) are summarised by eye (study eye and non study eye) and evaluation visit, and stratified by severity level.
  Only study eye's results are reported hereunder.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
letters
  Day 1 vs Day -15 | 0.7 (2.9) | 1.6 (5.8)
  Day 8 vs Day -15 | 0.5 (2.9) | 3.4 (6.3)
  Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Day 29 vs Day -15 | 1.3 (3.8) | 5.1 (11.7)
  Day 56 vs Day -15 | 1.2 (3.8) | 6.7 (10.6)

15. Secondary Outcome: Number of Participants With a Change in Fundus Ophthalmoscopy
Description: This test allows seeing inside the fundus of the eye and other structures using an ophthalmoscope. The fundus examination included assessments of vitreous, macula, retina and optic nerve head for both eyes. Only the results concerning the study eye are reported hereunder.
  These structures will be assessed according to the criteria outlined below.
  Vitreous The examiner will judge the appearance of the vitreous in the visual axis. Normal: Absence of any opacity Abnormal: Presence of opacity
  Macula, (Peripheral) Retina and Optic Nerve Head The examiner will provide a separate assessment of the macular, choroid and peripheral retina Normal: Absence of any structural or vascular change, inflammation, oedema or haemorrhage.
  Abnormal: Evidence of any ongoing or previous structural/vascular change, inflammation, oedema or haemorrhage.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
Participants
  Vitreous, Day 1 vs Day -15 | 0 | 0
  Vitreous, Day 8 vs Day -15 | 0 | 0
  Vitreous, Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Vitreous, Day 29 vs Day -15 | 0 | 0
  Vitreous, Day 56 vs Day -15 | 0 | 0
  Macula, Retina and Optic Nerve Head - Day 1 | 0 | 0
  Macula, Retina and Optic Nerve Head - Day 8 | 0 | 0
  Macula, Retina and Optic Nerve Head - Day 29: number analyzed (Participants) | 20 | 19
  Macula, Retina and Optic Nerve Head - Day 29 | 0 | 0
  Macula, Retina and Optic Nerve Head - Day 56 | 0 | 0

16. Secondary Outcome: Change From Baseline in Tear Film Osmolarity
Description: Values of tear film osmolarity and their changes from baseline (screening visit) are summarised by eye (study eye and non study eye) and evaluation visit and stratified by severity level. Only study eye's results are reported hereunder.
Time Frame: Changes from baseline up to day 56±4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
mOsm/L
  Day 1 vs Day -15 | -9.1 (13.1) | -0.8 (18.3)
  Day 8 vs Day -15 | -4.1 (16.2) | 0.5 (15.0)
  Day 29 vs Day -15: number analyzed (Participants) | 20 | 19
  Day 29 vs Day -15 | -5.5 (10.8) | -1.4 (19.0)
  Day 56 vs Day -15 | -4.8 (14.2) | 4.1 (19.8)

17. Secondary Outcome: Change From Baseline in Conjunctival Impression Cytology for Goblet Cells' Count
Description: Four conjunctival impression cytology samples (temporal, nasal, inferior and superior bulbar conjunctiva) for conjunctival goblet cell counts were performed in the worse eye (study eye).
  Conjunctival epithelium samples are obtained following the instillation of a preservative-free anaesthetic eye drop by slightly pressing on the bulbar conjunctiva a 0.1 μm cellulose acetate filter. When the disc is removed the apical layers of conjunctival epithelium remain "impressed" on it.
  Cells on the filter are fixed and stained. The final results will be expressed as mean ± SD of 3 consecutive optic fields for each sample.
  A higher number of goblet cells indicates a healthier eye.
Time Frame: Baseline, Day 1, Day 8, Day 29 and Day 56
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cell counts
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
cell counts
  Temporal Bulbar Conjunctiva, Day 1 vs Day -15: number analyzed (Participants) | 15 | 20
  Temporal Bulbar Conjunctiva, Day 1 vs Day -15 | -2.04 (7.66) | -0.19 (3.40)
  Temporal Bulbar Conjunctiva, Day 8 vs Day -15: number analyzed (Participants) | 17 | 19
  Temporal Bulbar Conjunctiva, Day 8 vs Day -15 | -2.25 (6.73) | 0.16 (2.19)
  Temporal Bulbar Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 15 | 18
  Temporal Bulbar Conjunctiva, Day 29 vs Day -15 | 0.03 (11.18) | 0.83 (2.72)
  Temporal Bulbar Conjunctiva, Day 56 vs Day -15: number analyzed (Participants) | 15 | 20
  Temporal Bulbar Conjunctiva, Day 56 vs Day -15 | -2.47 (7.86) | 0.00 (2.76)
  Nasal Bulbar Conjunctiva, Day 1 vs Day -15: number analyzed (Participants) | 15 | 19
  Nasal Bulbar Conjunctiva, Day 1 vs Day -15 | -0.84 (8.55) | -0.52 (2.50)
  Nasal Bulbar Conjunctiva, Day 8 vs Day -15: number analyzed (Participants) | 16 | 17
  Nasal Bulbar Conjunctiva, Day 8 vs Day -15 | 0.98 (14.02) | 1.24 (4.06)
  Nasal Bulbar Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 16 | 16
  Nasal Bulbar Conjunctiva, Day 29 vs Day -15 | 0.96 (9.14) | -0.06 (2.98)
  Nasal Bulbar Conjunctiva, Day 56 vs Day -15: number analyzed (Participants) | 17 | 16
  Nasal Bulbar Conjunctiva, Day 56 vs Day -15 | 0.99 (12.81) | 1.19 (3.89)
  Inferior Bulbar Conjunctiva, Day 1 vs Day -15: number analyzed (Participants) | 19 | 20
  Inferior Bulbar Conjunctiva, Day 1 vs Day -15 | -2.77 (7.49) | -2.17 (4.65)
  Inferior Bulbar Conjunctiva, Day 8 vs Day -15: number analyzed (Participants) | 19 | 19
  Inferior Bulbar Conjunctiva, Day 8 vs Day -15 | -1.11 (11.30) | -1.33 (3.41)
  Inferior Bulbar Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 19 | 19
  Inferior Bulbar Conjunctiva, Day 29 vs Day -15 | -3.79 (7.30) | -1.60 (3.11)
  Inferior Bulbar Conjunctiva, Day 56 vs Day -15: number analyzed (Participants) | 19 | 20
  Inferior Bulbar Conjunctiva, Day 56 vs Day -15 | -1.60 (8.94) | -1.07 (4.46)
  Superior Bulbar Conjunctiva, Day 1 vs Day -15: number analyzed (Participants) | 19 | 19
  Superior Bulbar Conjunctiva, Day 1 vs Day -15 | -2.28 (9.87) | 0.73 (2.23)
  Superior Bulbar Conjunctiva, Day 8 vs Day -15: number analyzed (Participants) | 18 | 18
  Superior Bulbar Conjunctiva, Day 8 vs Day -15 | -2.48 (12.53) | 0.33 (2.35)
  Superior Bulbar Conjunctiva, Day 29 vs Day -15: number analyzed (Participants) | 19 | 16
  Superior Bulbar Conjunctiva, Day 29 vs Day -15 | -4.44 (10.16) | 0.44 (1.93)
  Superior Bulbar Conjunctiva, Day 56 vs Day -15: number analyzed (Participants) | 18 | 18
  Superior Bulbar Conjunctiva, Day 56 vs Day -15 | -1.09 (10.45) | 1.07 (1.99)

18. Secondary Outcome: Mean Frequency of Artificial Tears Use
Description: During the treatment with rhNGF at both doses (from day 1 to day 29), and in the follow-up period (from day 29 to day 56) the mean frequency of daily use of artificial tears was measured.
Time Frame: Day 1-Day 8, Day 9-Day 29, Day 30-Day 56 intervals
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: uses per day
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
Number analyzed (Participants) | 20 | 20
uses per day
  Day 1-Day 8: number analyzed (Participants) | 10 | 12
  Day 1-Day 8 | 1.813 (1.894) | 1.083 (1.541)
  Day 9-Day 29: number analyzed (Participants) | 10 | 13
  Day 9-Day 29 | 2.133 (2.814) | 1.271 (1.334)
  Day 30-Day 56: number analyzed (Participants) | 11 | 12
  Day 30-Day 56 | 2.869 (2.961) | 2.460 (2.860)

ADVERSE EVENTS:
Time Frame: From screening throughout the study until the final visit, up to 56 days
Description: More specifically, adverse events are assessed at screening (visit 1), at visits 2-6 and at visit 7 (final visit, Day 56)
Arm/Group | Group 1 - rhNGF 20 μg/mL | Group 2 - rhNGF 4 μg/mL
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 14/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - rhNGF 20 μg/mL (N=20) | Group 2 - rhNGF 4 μg/mL (N=20)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - rhNGF 20 μg/mL (N=20) | Group 2 - rhNGF 4 μg/mL (N=20)
Abnormal sensation in eye (Eye disorders) | 4 (4) | 8 (9)
Eye pain (Eye disorders) | 5 (7) | 6 (7)
Eye irritation (Eye disorders) | 3 (6) | 7 (7)
Eye pruritus (Eye disorders) | 2 (4) | 5 (5)
Vision blurred (Eye disorders) | 3 (4) | 2 (2)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 4 (4)
Photophobia (Eye disorders) | 1 (2) | 3 (3)
Lacrimation increased (Eye disorders) | 0 (0) | 3 (3)
Visual impairment (Eye disorders) | 1 (1) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid sensory disorder (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Vitrous detachment (Eye disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
LImitations and caveats non specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No